CLINICAL TRIAL: NCT06738732
Title: Preliminary Evaluation of the Safety and Efficacy of CBD Delivery with the A-Synaptic GT4 Transdermal Delivery System in Individuals Diagnosed with Dravet Syndrome And/or Lennox-Gastaut Syndrome
Brief Title: CBD Delivery with the A-Synaptic GT4 Transdermal Delivery System in with Dravet Syndrome And/or Lennox-Gastaut Syndrome
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexander Rotenberg (Other)
Collaborators: A-Synaptic (Unknown)
Responsible Party: Sponsor-Investigator, Alexander Rotenberg, Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00047233
Record Dates: First submitted 2024-11-08; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Lennox-Gastaut Syndrome (LGS); Dravet Syndrome (DS)
Keywords: CBD; transdermal
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsies, Myoclonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active Therapy (Experimental): CBD: GT4 Transdermal Delivery System
  Interventions: Drug: CBD: GT4 Transdermal Delivery System

INTERVENTIONS:
Drug: CBD: GT4 Transdermal Delivery System — CBD: GT4 Transdermal Delivery System

SUMMARY:
This study is a preliminary open-label, single-arm Phase II investigation into the safety and efficacy of transdermal cannabidiol (CBD) delivered using GT4 skin bream technology in individuals diagnosed with Dravet and/or Lennox-Gastatu syndrome (DS and/or LGS). We aim to enroll 25 participants between the ages of 2 and 55 diagnosed with DS and/or LGS.

Transdermal delivery of cannabinoids may provide advantages over other traditional routes of administration. Noted advantages include avoidance of first pass metabolism which mitigates potentially dangerous drug-drug interactions due to delayed cannabinoid accumulation, and more stable and constant plasma cannabinoid concentrations. GT4 technology, uses emulsion technology containing penetrating agents, basement membrane disruptors, and vasodilators to overcome hydrophilic and lipophilic structures to open channels and transport cannabinoids deep into the dermis layer of the skin. Once in the dermis, vasodilators dilate the capillary bed to increase fluid dynamic flow into and out of the application site, delivering cannabinoids into the blood stream.

The primary objective is to investigate the safety and efficacy of CBD delivery with the A-Synaptic GT4 Transdermal Delivery System in individuals diagnosed with DS and/orLGS. Dr. Rotenberg will apply for and hold the expanded access IND for this study, as the sponsor is running this study as an investigator-initiated study.

The study consists of 11 visits over ~160 days, dosing begins at Visit #2.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the age of 2-55 years, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation), have been post-menopausal for at least 1 year prior to screening, or have not reached menarche Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active
3. Clinically confirmed and documented diagnosis of refractory DS and/or LGS. Documentation of diagnosis must be provided by a neurologist, pediatrician, or primary care practitioner
4. Reported ≥4 countable seizures during the 28-day run in period
5. Participants taking ≥1 AED at a stable dose for ≥4 weeks prior to screening, and participants and/or caregivers willing to maintain dose for duration of study period
6. Non-pharmacological therapies (e.g., vagus nerve stimulation, ketogenic diet, modified Atkins diet) stable for ≥4 weeks prior to screening, and participants and/or caregivers willing to maintain a stable regimen for the duration of the study period
7. Adults to provide voluntary, written, informed consent to participate in the study. If under the age of consent or unable to consent due to cognitive impairment, the participant and the participant's parent(s), legal guardian(s), or caregiver(s) to provide voluntary, written, informed assent and consent, respectively, for participation in the study
8. Otherwise healthy as determined by medical history, laboratory results, electroencephalogram (EEG), vital signs, and physical examination, as assessed by the QI/MD

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product's active and/or inactive ingredients
3. Acute or chronic skin disease (e.g., atopic dermatitis, eczema, rosacea, psoriasis) or dermatological conditions (scars, moles, etc.) in the proposed area of application that may interfere with the application and absorption of the investigational product, as assessed by the QI/MD
4. Etiology of participant seizures is related to progressive neurologic disease, as assessed by the QI/MD.
5. Currently prescribed >4 concurrent AEDs
6. Current unstable significant psychiatric or psychological condition (e.g., schizophrenia, bipolar disorder, clinical depression, eating disorders) and/or history of suicidal behavior or any suicidal ideation as assessed by the C-SSRS at screening, as appropriate, as assessed by the QI/MD (See Section 9.13.2)
7. History of psychosis in immediate family including schizophrenia and affective psychosis
8. Anoxic episode requiring resuscitation in the past 6 months
9. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI/MD
10. Type I or Type II diabetes
11. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI/MD on a case-by-case basis
12. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI/MD on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
13. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI/MD
14. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI/MD
15. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
16. Individuals with an autoimmune disease or are immune compromised
17. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis
18. Self-reported confirmation of blood/bleeding disorders as assessed by QI/MD
19. Use of medical or recreational cannabinoid products prior to screening (see Section 7.3). Participants must agree to abstain for the duration of the run-in and study period
20. Regular use of tobacco or nicotine products in the past 6 months and during the run-in and study period, as assessed by the QI/MD
21. Alcohol intake average of >2 standard drinks per day, as assessed by the QI/MD. Occasional consumers required to abstain for the duration of the run-in and study period
22. Alcohol or drug abuse within the last 24 months
23. Current use of any prescribed or over-the counter medications and/or supplements that may affect the safety and/or efficacy of the investigational product, as assessed by the QI/MD (See Sections 7.3.1 and 7.3.2)
24. Plans to travel outside country of residence during the study period
25. Clinically significant abnormal laboratory results, adverse events, or abnormalities in the EEG at screening, as assessed by the QI/MD
26. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI/MD
27. Any other condition, chronic disease, or lifestyle factor, that, in the opinion of the QI/MD, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 2 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Compliance | 112 Days
  Proportion of participants compliant with study dosing regimen for visits at baseline, 7, 14, 21, 28, 56, 84, and 112 days post treatment;
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 112 Days
  Pre-emergent and post-emergent adverse events will be described in separate frequency tables. The description, frequency, type, severity, causality, and outcome of each adverse event will also be listed.

SECONDARY OUTCOMES:
Seizure Frequency | 112 Days
  Proportion, relative to baseline will be computed for three seizure types: (1) drop, (2) generalized tonic, and (3) generalized tonic-clonic. Seizure freqeuncy values will be collected 28, 56, 84 and 112 days post treatment to compute percent change in frequency at 28, 56, 84 and 112 days post treatment.
CBD, 7-COOH-CBD, and 7-OH-CBD blood concentrations, and blood concentrations of concomitant AEDs | 112 Days
  Blood will be collected at morning trough, before morning medicaiton adminitration. Summary statistics including means, standard deviations, medians, minimums, maximums, on secondary outcome variables: CBD, 7-COOH-CBD, and 7-OH-CBD blood concentrations, and blood concentrations of concomitant AEDs will be obtained for baseline, 1, 7, 14, 21, 28, 56, 84 and 112 days post treatment for the overall ITT and PP populations. Similar summary statistics will also be obtained for changes from baseline to 1, 7, 14, 21, 28, 56, 84 and 112 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rotenberg, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Childrens' Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No